CLINICAL TRIAL: NCT01025752
Title: IVR-based Cognitive Behavior Therapy for Chronic Low Back
Brief Title: Interactive Voice Response (IVR)-Based Treatment for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 09-058
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2017-10

CONDITIONS: Chronic Low Back Pain
Keywords: chronic pain; cognitive behavior therapy; low back pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Ten session IVR-based cognitive behavior therapy intervention for chronic low back pain
  Interventions: Behavioral: IVR based cognitive behavioral therapy
- Arm 2 (Active Comparator): Ten session face to face cognitive behavior therapy for chronic low back pain
  Interventions: Behavioral: Face to face cognitive behavior therapy

INTERVENTIONS:
Behavioral: Face to face cognitive behavior therapy — Ten session face to face cognitive behavior therapy for chronic low back pain
  Arms: Arm 2
Behavioral: IVR based cognitive behavioral therapy — Ten session cognitive behavior therapy for chronic low back pain using interactive voice response therapy
  Arms: Arm 1

SUMMARY:
The proposed study will test how well an innovative method, interactive voice response (IVR), can be used for delivering an treatment for chronic low back pain. The use of IVR will improve the accessibility of treatment to Veterans. IVR is a computerized interface that allows patients to use their telephone to: 1) obtain pre-recorded didactic information, 2) report data regarding pain-related symptoms and adherence to pain coping skill practice, and 3) receive personalized therapist feedback. Although CBT has been shown to be effective in reducing pain intensity, traditional CBT requires patients to make frequent office visits. The use of IVR will allow Veterans to access CBT from their home via a touch-tone telephone, thereby allowing them to access treatment at their convenience without travel to the VA for an outpatient appointment. Veterans with chronic low back pain will be randomized in equal numbers to receive either standard CBT or IVR-based CBT. Veterans in both conditions will receive 10 session of treatment designed to help them manage their chronic pain using pain coping skills. The primary outcome measure will be pain intensity.

DETAILED DESCRIPTION:
OBJECTIVES: The primary purpose of this study is to test the efficacy of an innovative method, interactive voice response (IVR), for delivering an empirically validated psychological (cognitive behavior therapy [CBT]) treatment for chronic pain in order to improve access and sustainability of this intervention. The primary clinical equivalence hypothesis states that Veterans with chronic low back pain (CLBP) receiving IVR-based CBT (ICBT) will demonstrate, relative to standard face-to-face CBT (CBT), equivalent declines in reports of pain intensity as measured by the numeric rating scale at post-treatment and follow-up. The secondary hypothesis states that Veterans with CLBP receiving ICBT, relative to CBT, will demonstrate equivalent declines in reports of pain-related interference and emotional distress at post-treatment and follow-up.

RESEARCH DESIGN: A randomized design will be employed in which standard CBT (CBT) is compared to an Interactive CBT (ICBT) treatment condition. Participants will be randomized in equal numbers to both conditions. Repeated assessments of key outcome domains will occur at pretreatment/baseline and at 3 and 6 months following baseline.

METHODOLOGY: Subjects will be 230 patients receiving care at the VA Connecticut Healthcare System who report chronic low back pain. The primary criteria for inclusion are constant pain of at least three months duration with at least a moderate level of average pain (i.e., scores of 4 or greater on a 0 (no pain) to 10 (worst pain imaginable) on a numerical rating scale of average pain. All patients must have access to a touch-tone telephone. Excluded will be patients with life threatening or acute physical illness, current alcohol or substance abuse or dependence, current psychosis, suicidal ideation, dementia, and individuals seeking surgical pain treatment. Comprehensive evaluations will be conducted at each assessment interval. Following completion of written consent and an initial baseline evaluation, participants will be randomized to one of the two treatments. Sessions will be audiotaped to ensure the fidelity of the face-to-face CBT sessions and the personalized therapist feedback in the IVR-based CBT condition. Both conditions will involve 10 outpatient therapy sessions with a psychologist trained experienced in the delivery of these treatments. Adherence to coping skill practice will be assessed using IVR for both treatment groups. Analysis of primary and secondary outcome measures will employ mixed-effects models, which will account for the clustering induced by repeated measures on individual patients.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least a moderate level of pain (i.e., pain scores of > or = 4) and presence of pain for a period of > or = 3 months
* ability to participate safely in the walking portion of the intervention as evidenced by ability to walk at least one block
* availability of a touch-tone telephone and computer with internet access in the participant's residence
* Veteran receiving care at VA Connecticut Healthcare System

Exclusion Criteria:

* life threatening or acute medical condition that could impair participation (e.g., severe chronic obstructive pulmonary disease, lower limb amputation, terminal cancer);
* psychiatric condition (e.g., active substance abuse, psychosis or suicidality) that could impair participation
* surgical interventions for pain during their participation in this study
* sensory deficits that would impair participation (e.g., hearing loss to a degree that telephone usage is not possible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2011-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia A. Heapy, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Heapy AA, Higgins DM, LaChappelle KM, Kirlin J, Goulet JL, Czlapinski RA, Buta E, Piette JD, Krein SL, Richardson CR, Kerns RD. Cooperative pain education and self-management (COPES): study design and protocol of a randomized non-inferiority trial of an interactive voice response-based self-management intervention for chronic low back pain. BMC Musculoskelet Disord. 2016 Feb 16;17:85. doi: 10.1186/s12891-016-0924-z. PMID 26879051
- [Derived] MacLean RR, Buta E, Higgins DM, Driscoll MA, Edmond SN, LaChappelle KM, Ankawi B, Krein SL, Piette JD, Heapy AA. Using Daily Ratings to Examine Treatment Dose and Response in Cognitive Behavioral Therapy for Chronic Pain: A Secondary Analysis of the Co-Operative Pain Education and Self-Management Clinical Trial. Pain Med. 2023 Jul 5;24(7):846-854. doi: 10.1093/pm/pnac192. PMID 36484691
- [Derived] Heapy AA, Tankha H, Higgins DM, Driscoll M, LaChappelle KM, Goulet JL, Buta E, Piette JD, Kerns RD, Krein SL. Incorporating walking into cognitive behavioral therapy for chronic pain: safety and effectiveness of a personalized walking intervention. J Behav Med. 2021 Apr;44(2):260-269. doi: 10.1007/s10865-020-00193-8. Epub 2021 Jan 1. PMID 33386530
- [Derived] Heapy AA, Higgins DM, Goulet JL, LaChappelle KM, Driscoll MA, Czlapinski RA, Buta E, Piette JD, Krein SL, Kerns RD. Interactive Voice Response-Based Self-management for Chronic Back Pain: The COPES Noninferiority Randomized Trial. JAMA Intern Med. 2017 Jun 1;177(6):765-773. doi: 10.1001/jamainternmed.2017.0223. PMID 28384682

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans with chronic back pain from VA Connecticut Healthcare System and surrounding community areas were recruited from June 2012-July 2015.
Pre-assignment Details: Eligibility screening was conducted by the research assistant via interview and medical record review. Participants who enrolled then subsequently found ineligible from further baseline assessment questionnaires were not randomized to a treatment arm, and excluded from the study (i.e. substance abuse, severe depression, cognitive impairment), n=9.
Groups:
- Arm 1: IVR CBT: Ten session IVR-based cognitive behavior therapy for chronic low back pain
  IVR based cognitive behavioral therapy: Ten session cognitive behavior therapy for chronic low back pain using interactive voice response therapy
- Arm 2: F2F CBT: Ten session face to face cognitive behavior therapy for chronic low back pain
  Face to face cognitive behavior therapy: Ten session face to face cognitive behavior therapy for chronic low back pain
Period: Overall Study
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Started | 62 | 63
Completed | 54 | 50
Not Completed | 8 | 13
Not completed — Lost to Follow-up | 7 | 10
Not completed — Physician Decision | 1 | 3

BASELINE CHARACTERISTICS:
Population: 134 participants were consented, 9 failed baseline screening measures and 125 were randomized to either IVR CBT or F2F CBT.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.8) | 56.7 (11.5) | 57.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 49 | 48 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Balck, not Hispanic | 14 | 18 | 32
  Hispanic | 3 | 6 | 9
  White, not Hispanic | 43 | 37 | 80
  Other | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 63 | 125

OUTCOME MEASURES:

1. Primary Outcome: Change in Numeric Rating Scale of Pain Intensity
Description: An 11-point NRS for pain was administered to patients, with 0 representing "No Pain" and 10 representing "Worst Possible Pain." Patients were asked to rate the level of pain that best represented their experience of worst pain, least pain and average pain over the past week. We computed the change from baseline.
Time Frame: post-treatment (12 weeks), 3 and 6 months post-baseline
Population: The number analyzed in rows differs because we analyzed the available follow-up questionnaire data for each participant (some participants did not complete the questionnaires at all time points).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Number analyzed (Participants) | 54 | 50
units on a scale
  post-treatment (12 weeks): number analyzed (Participants) | 52 | 42
  post-treatment (12 weeks) | -0.77 [-1.29 to -0.26] | -0.84 [-1.39 to -0.29]
  3 months post-baseline: number analyzed (Participants) | 49 | 45
  3 months post-baseline | -1.23 [-1.73 to -0.72] | -1.00 [-1.52 to -0.48]
  6 months post-baseline: number analyzed (Participants) | 49 | 45
  6 months post-baseline | -0.51 [-1.06 to 0.04] | -0.44 [-1.01 to 0.14]
Statistical Analysis 1: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; post-treatment (12 weeks) time point; Test type: Non-Inferiority — A 20% (1.4) reduction in NRS for pain intensity from baseline was considered minimally clinically important the non-inferiority margin was set at one NRS unit. The required sample size was 230 participants. Because enrollment was slower than expected and the standard deviation in the primary outcome was less than the initial power calculation (1.6 vs. 2.45) we conducted a sample size recalculation, based on observed data to determine that we would need 42 completers per arm for 80% power; p = 0.007, Mixed Models Analysis — Non-inferiority margin of 1; The models includes treatment arm, time, treatment-by-time interaction, baseline NRS, stratification variables (distance from VA & back pain cause); Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.67 to 0.80] — The upper limit (0.80) fell below the non-inferiority margin of 1
Statistical Analysis 2: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 3 month post-baseline time point; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Mixed Models Analysis — Non-inferiority margin of 1; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.94 to 0.49] — The upper limit (0.49) fell below the non-inferiority margin of 1
Statistical Analysis 3: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 6 month post- baseline time point; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.004, Mixed Models Analysis — The non-inferiority margin is 1; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.86 to 0.71] — The upper limit (0.71) fell below the non-inferiority margin of 1

2. Secondary Outcome: Change in Multidimensional Pain Inventory Interference Subscale
Description: The interference subscale of the West Haven-Yale Multidimensional Pain Inventory (WHYMPI) assesses pain-related interference with quality of life. Scores ranging from 0-6, with higher scores indicating more interference. We computed the change from baseline.
Time Frame: post-treatment (12 weeks), 3 and 6 months post-baseline
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Number analyzed (Participants) | 53 | 51
units on a scale
  post-treatment (12 weeks): number analyzed (Participants) | 51 | 43
  post-treatment (12 weeks) | -0.37 [-0.66 to -0.08] | -0.04 [-0.35 to 0.26]
  3 months post-baseline: number analyzed (Participants) | 48 | 46
  3 months post-baseline | -0.37 [-0.73 to 0.00] | -0.02 [-0.40 to 0.35]
  6 months post-baseline: number analyzed (Participants) | 48 | 45
  6 months post-baseline | -0.12 [-0.50 to 0.26] | -0.09 [-0.48 to 0.30]
Statistical Analysis 1: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; Post-treatment (12 weeks) time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.74 to 0.09]
Statistical Analysis 2: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 3 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.20, Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.87 to 0.18]
Statistical Analysis 3: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 6 months post baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.93, Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.57 to 0.52]

3. Secondary Outcome: Change in Roland Morris Disability Questionnaire
Description: The RMDQ (Roland & Morris, 1983) is a 24-item checklist designed for patients to identify the level of disability and functional status associated with chronic low back pain. Patients are instructed to endorse items that describe their functional status that day. Scores range from 0-24, with higher scores indicating more disability. We computed the change from baseline.
Time Frame: post-treatment (12 weeks), 3 and 6 months post-baseline
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Number analyzed (Participants) | 53 | 51
units on a scale
  post-treatment (12 weeks): number analyzed (Participants) | 51 | 43
  post-treatment (12 weeks) | -2.92 [-4.16 to -1.69] | -2.42 [-3.74 to -1.11]
  3 months post-baseline: number analyzed (Participants) | 48 | 46
  3 months post-baseline | -3.38 [-4.75 to -2.02] | -1.86 [-3.25 to -0.46]
  6 months post-baseline: number analyzed (Participants) | 48 | 45
  6 months post-baseline | -2.63 [-3.90 to -1.35] | -2.02 [-3.32 to -0.71]
Statistical Analysis 1: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; post-treatment (12 weeks) time point; Test type: Other; p = 0.58, Mixed Models Analysis; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-2.29 to 1.29]
Statistical Analysis 2: Comparison: Arm 1: IVR CBT; 3 months post-baseline time point; Test type: Other; p = 0.12, Mixed Models Analysis; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-3.46 to 0.41]
Statistical Analysis 3: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 6 months post-baseline time point; Test type: Other; p = 0.51, Mixed Models Analysis; Mean Difference (Final Values) = -0.61, 95% CI 2-sided [-2.42 to 1.20]

4. Secondary Outcome: Change in Veterans Short Form-36 Health Status Questionnaire: Physical Component Scale
Description: The SF-36V is an adaptation of the Medical Outcomes Study SF-36 (Ware & Sherbourne, 1992) intended to apply to veteran-specific health-related quality of life. The SF-36 can also be divided into two aggregate summary measures the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The lower the score, the more disability, range 0-100. We computed the change from baseline.
Time Frame: post-treatment (12 weeks), 3 and 6 months post-baseline
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Number analyzed (Participants) | 52 | 48
units on a scale
  post-treatment (12 weeks): number analyzed (Participants) | 47 | 40
  post-treatment (12 weeks) | 2.20 [0.43 to 3.96] | 1.91 [0.01 to 3.81]
  3 months post-baseline: number analyzed (Participants) | 45 | 42
  3 months post-baseline | 2.05 [0.09 to 4.02] | 0.90 [-1.15 to 2.95]
  6 months post-baseline: number analyzed (Participants) | 45 | 41
  6 months post-baseline | 1.50 [-0.44 to 3.45] | 2.09 [0.03 to 4.14]
Statistical Analysis 1: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; post-treatment (12 weeks) time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.83, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-2.30 to 2.87]
Statistical Analysis 2: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 3 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.42, Mixed Models Analysis; Mean Difference (Final Values) = 1.15, 95% CI 2-sided [-1.68 to 3.98]
Statistical Analysis 3: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 6 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.68, Mixed Models Analysis; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-3.40 to 2.24]

5. Secondary Outcome: Change in Veterans Short Form-36 Health Status Questionnaire: Mental Component Scale
Description: as for outcome 4
Time Frame: post-treatment (12 weeks), 3 and 6 months post-baseline
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Number analyzed (Participants) | 52 | 48
units on a scale
  post-treatment (12 weeks): number analyzed (Participants) | 47 | 40
  post-treatment (12 weeks) | 1.67 [-0.36 to 3.71] | 0.42 [-1.74 to 2.59]
  3 months post-baseline: number analyzed (Participants) | 45 | 42
  3 months post-baseline | 1.39 [-0.86 to 3.64] | 1.01 [-1.33 to 3.35]
  6 months post-baseline: number analyzed (Participants) | 45 | 41
  6 months post-baseline | 0.96 [-1.41 to 3.33] | -1.47 [-3.96 to 1.02]
Statistical Analysis 1: Comparison: Arm 1: IVR CBT; post-treatment (12 weeks) time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.40, Mixed Models Analysis; Mean Difference (Final Values) = 1.25, 95% CI 2-sided [-1.66 to 4.16]
Statistical Analysis 2: Comparison: Arm 1: IVR CBT; 3 months post-baseline. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.81, Mixed Models Analysis; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-2.82 to 3.58]
Statistical Analysis 3: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 6 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.16, Mixed Models Analysis; Mean Difference (Final Values) = 2.43, 95% CI 2-sided [-0.96 to 5.82]

6. Secondary Outcome: Change in Beck Depression Inventory-II
Description: Depressive symptom severity was assessed using the BDI-II, higher scores indicate more depressive symptomology, range 0-63. We computed the change from baseline.
Time Frame: post-treatment (12 weeks), 3 and 6 months post-baseline
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Number analyzed (Participants) | 54 | 51
units on a scale
  post-treatment (12 weeks): number analyzed (Participants) | 52 | 43
  post-treatment (12 weeks) | -1.00 [-2.79 to 0.78] | -1.25 [-3.14 to 0.65]
  3 months post-baseline: number analyzed (Participants) | 49 | 46
  3 months post-baseline | -0.49 [-2.61 to 1.64] | 0.78 [-1.40 to 2.96]
  6 months post-baseline: number analyzed (Participants) | 49 | 45
  6 months post-baseline | 0.89 [-1.62 to 3.40] | 1.62 [-0.97 to 4.21]
Statistical Analysis 1: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; post-treatment (12 weeks time point). (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.85, Mixed Models Analysis; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-2.32 to 2.80]
Statistical Analysis 2: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 3 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.40, Mixed Models Analysis; Mean Difference (Final Values) = -1.27, 95% CI 2-sided [-4.27 to 1.73]
Statistical Analysis 3: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 6 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.68, Mixed Models Analysis; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-4.30 to 2.83]

7. Secondary Outcome: Change in Pittsburgh Sleep Quality Index
Description: The PSQI assess sleep quality, with lower scores indicating better sleep, range 0 to 21.We computed the change from baseline.
Time Frame: post-treatment (12 weeks), 3 and 6 months post-baseline
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Number analyzed (Participants) | 48 | 49
units on a scale
  post-treatment (12 weeks): number analyzed (Participants) | 47 | 38
  post-treatment (12 weeks) | -2.03 [-2.94 to -1.12] | -1.09 [-2.06 to -0.11]
  3 months post-baseline: number analyzed (Participants) | 45 | 42
  3 months post-baseline | -1.33 [-2.21 to -0.44] | -1.21 [-2.12 to -0.29]
  6 months post-baseline: number analyzed (Participants) | 44 | 42
  6 months post-baseline | -0.87 [-1.99 to 0.24] | -1.25 [-2.38 to -0.11]
Statistical Analysis 1: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; post-treatment (12 weeks) time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.17, Mixed Models Analysis; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-2.28 to 0.40]
Statistical Analysis 2: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 3 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.86, Mixed Models Analysis; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-1.39 to 1.16]
Statistical Analysis 3: Comparison: Arm 1: IVR CBT vs Arm 2: F2F CBT; 6 months post-baseline time point. (Mean difference of IVR CBT- F2F CBT); Test type: Other; p = 0.64, Mixed Models Analysis; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-1.22 to 1.97]

ADVERSE EVENTS:
Arm/Group | Arm 1: IVR CBT | Arm 2: F2F CBT
Serious Adverse Events (participants affected / at risk) | 1/62 | 1/63
Other Adverse Events (participants affected / at risk) | 14/62 | 19/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: IVR CBT (N=62) | Arm 2: F2F CBT (N=63)
Infection of foot lesion (Infections and infestations) | 0 (0) | 1 (1) — Unrelated to study
Cardiac disorder event (Cardiac disorders) | 1 (1) | 0 (0) — Unrelated to study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: IVR CBT (N=62) | Arm 2: F2F CBT (N=63)
Trip or Fall (General disorders) | 5 (5) | 6 (7)
Muscle or joint pain increase (General disorders) | 11 (19) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No